CLINICAL TRIAL: NCT05594368
Title: Dose Escalation for Stereotactic Cardiac Radiation Therapy of Recurrent Ventricular Tachyarrhythmia - a Multi Center, Phase II Clinical Trial
Brief Title: Dose Escalation for SBRT of Recurrent VT Ventricular Tachyarrhythmia - a Single Center, Phase II Clinical Trial
Acronym: DEFT STAR
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022-00262
Record Dates: First submitted 2022-10-21; First posted 2022-10-26 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2025-02

CONDITIONS: Ventricular Tachycardia
MeSH Terms: conditions — Tachycardia, Ventricular

STUDY DESIGN:
Intervention Model Description: The study is designed as a one arm, multi-center dose escalation trial employing the i3+3 design.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Dose escalating stereotactic arrhythmia radioablation to treat ventricular tachycardia (VT) (Experimental)
  Interventions: Device: Dose escalating stereotactic arrhythmia radioablation to treat ventricular tachycardia (VT)

INTERVENTIONS:
Device: Dose escalating stereotactic arrhythmia radioablation to treat ventricular tachycardia (VT) — Dose escalating stereotactic arrhythmia radioablation to treat ventricular tachycardia (VT) refractory to conventional antiarrhythmic and catheter ablation-based therapy. First patients will be treated with a dose from 25 Gy prescribed to the 65-90% target volume encompassing isodose escalating to a maximum of 32.5 Gy prescribed to the 65-90% isodose.

SUMMARY:
The objective of this study is to demonstrate that higher radiation doses are necessary to induce transmural scar formation which is currently assumed to be the underlying mechanism of successful long-term efficacy of VT treatment and therefore dose-escalation will lead to a significantly reduced long-term VT recurrence rate compared to the currently applied single dose of 25 Gy.

ELIGIBILITY:
Inclusion Criteria:

Patients with structural heart disease, in particular ischemic and non-ischemic cardiomyopathy: Implanted ICD and/or CRT-D. Prior ≥1 failed catheter ablation (with endocardial ± epicardial approach based on the substrate location and the ECG morphology of clinical VTs) procedure to control sustained monomorphic VT using currently recommended mapping and ablation techniques,2 or patients in whom ablation is not feasible. Reasons for lack of epicardial ablation and non-feasibility of catheter ablation must be specified. Sustained VT recurrence after catheter ablation on optimised antiarrhythmic medication.

Age ≥18 years. IRB-approved, written informed consent must be provided

Exclusion Criteria:

Patients with only premature ventricular contractions.

Patients with sustained VT/VF who demonstrate:

Acute myocardial infarction; Primary electrical disease (channelopathy); Reversible and treatable cause (e.g., drug-induced or intoxication) of VT that can be adequately addressed otherwise; A target that cannot be safely and precisely defined based on stereotactic radiotherapy accuracy requirements (e.g., anatomical interference from OARs, overlapping prior radiation therapy to the thoracic region); Pregnancy or breastfeeding; Inability to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
safety measured by registered radiation associated adverse events up to 90 days | up to 90 days
  safety measured by registered radiation associated adverse events

SECONDARY OUTCOMES:
Radiation associated serious adverse event (at least grade 4 or 5 according to CTCAE v5) | As assessed at 90 days

CONTACTS AND LOCATIONS:
Locations (2):
- University Hospital Ostrava, Ostrava, Czechia
- University Hospital Zurich, Zurich, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Kovacs B, Mayinger M, Ehrbar S, Fesslmeier D, Ahmadsei M, Sazgary L, Manka R, Alkadhi H, Ruschitzka F, Duru F, Papachristofilou A, Sticherling C, Blamek S, Golba KS, Guckenberger M, Saguner AM, Andratschke N. Dose escalation for stereotactic arrhythmia radioablation of recurrent ventricular tachyarrhythmia - a phase II clinical trial. Radiat Oncol. 2023 Nov 8;18(1):185. doi: 10.1186/s13014-023-02361-x. PMID 37941012